CLINICAL TRIAL: NCT03055117
Title: Individual Versus Group-based Exercise Rehabilitation for Shoulder Disorders
Brief Title: Individual Versus Group-based Exercise Rehabilitation for Shoulder Disorders: a Randomised Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regional Hospital West Jutland (Other)
Collaborators: University of Aarhus (Other); Central Denmark Region (Other)
Responsible Party: Principal Investigator, David H Christiansen, Researcher, Regional Hospital West Jutland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1-10-72-178-16
Record Dates: First submitted 2017-02-03; First posted 2017-02-16 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Shoulder Pain
Keywords: Shoulder pain; Physiotherapy; Rehabilitation; Exercise
MeSH Terms: conditions — Shoulder Pain; Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group-based exercise rehabilitation (Experimental): Group-based rehabilitation: Group-based sessions (4-8 patients per group) with physiotherapist and home training for 8 weeks (maximum of 12 training sessions).
  Interventions: Behavioral: Group-based exercise rehabilitation; Behavioral: Home exercise
- Individual exercise rehabilitation (Active Comparator): Individual rehabilitation: One-on-one sessions with physiotherapist and home training for 8 weeks (maximum of 12 training sessions).
  Interventions: Behavioral: Individual exercise rehabilitation; Behavioral: Home exercise
- Home exercise (Active Comparator): Home exercise: Instruction in home exercise by physiotherapist, with maximum of 4 follow-up consultations over a period of 8 weeks.
  Interventions: Behavioral: Home exercise

INTERVENTIONS:
Behavioral: Group-based exercise rehabilitation — Group- based physiotherapy-led exercise rehabilitation
  Arms: Group-based exercise rehabilitation
Behavioral: Individual exercise rehabilitation — Individual physiotherapy-led exercise rehabilitation
  Arms: Individual exercise rehabilitation
Behavioral: Home exercise — Supervised home exercise

SUMMARY:
Degenerative shoulder disorders are frequent in the Danish population and often cause disability and sick leave. After hospital discharge patients are often referred to physiotherapy rehabilitation as part of the treatment, and it is often assumed that one-on-one sessions will yield better results than group-based sessions, because individual needs can be better meet and targeted

The project aims to evaluate the effect and cost-effectiveness of group- based exercise rehabilitation as compared to individual exercise rehabilitation in patients with degenerative shoulder disorders.

.

DETAILED DESCRIPTION:
The study is a three-armed controlled randomized trial in which a total of 180 patients referred to the municipal rehabilitation after hospital treatment due to shoulder disorders in 6 municipalities in Region Midtjylland expected to participate. Patients will be allocated to either 1) Group-based rehabilitation 2) Individual rehabilitation or 3) Home exercise.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and above, ability to speak and understand Danish and referred to physiotherapy rehabilitation after hospital conservative or surgical treatment under diagnose of rotator cuff/shoulder impingement or acromioclavicular osteoarthritis (International Classification of Diseases 10th revision [ICD-10] group M75.1-M75.8, M19.8).

Exclusion Criteria:

* Influence of co-morbidity, psychiatric illness, pregnancy, fullthickness rotator cuff tear, rotator cuff repair surgery, traumatic lesion, rheumatoid arthritis, frozen shoulder, glenohumeral osteoarthritis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2017-02-16 (Actual); Primary Completion 2018-08-27 (Actual); Study Completion 2018-08-27 (Actual)

PRIMARY OUTCOMES:
Disability wil be assessed by The Disabilities of the Arm, Shoulder and Hand questionnaire - shortened version (Quick DASH) | 6 monhts
  Sum score 0-100

SECONDARY OUTCOMES:
Cost-effectiveness across study arms measured by the EuroQol (EQ-5D) questionnaire | 6 months
  Quality of life scale EQ-5D-5L will be used to calculate quality adjusted life years (QALYs) used in the health economic evaluation
Time off work (weeks) assessed by the Danish Register of Sickness absence compensation benefits and Social transfer payments | 6 months
  Register
Pain intensity | 6 months
  Numeric scale (0-10)
Patients impression of change of overall shoulder condition | 6 months
  Single item question
Patient Acceptable Symptom State (PASS) | 6 months
  Single item question. The highest level of symptom at which patients find their condition acceptable
Well-being wil be assessed by the WHO-5 Well-being Index questionnaire | 6 months
  Sum score of 5 items 0-100
Re-presentations after discharge from rehabilitation will be obtained by Danish National Rehabilitation | 6 months
  Register number of contacts
Fear avoidance Beliefs and risk of chronicity the Orebro Musculoskeletal Pain Screening Questionnaire | 6 months
  Sumscore 0-20
Confidence will be assessed by one item from the Danish Cancer Society PREM (Barometer) Questionnaire | 3 months
  Single item question.
Safety will be assessed by one item from the Danish Cancer Society PREM (Barometer) Questionnaire | 3 months
  Single item question.
Satisfaction will be assessed by one item from the Danish Cancer Society PREM (Barometer) Questionnaire | 3 months
  Single item question.

CONTACTS AND LOCATIONS:
Overall Officials: David H Christiansen, PhD, Principal Investigator — Occupational Medicine Regional Hospital West Jutland University Research Clinic
Locations (1):
- David H Christiansen, Herning, Central Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Christiansen DH, Hjort J. Group-based exercise, individually supervised exercise and home-based exercise have similar clinical effects and cost-effectiveness in people with subacromial pain: a randomised trial. J Physiother. 2021 Apr;67(2):124-131. doi: 10.1016/j.jphys.2021.02.015. Epub 2021 Mar 17. PMID 33744191